CLINICAL TRIAL: NCT00080756
Title: Biomarkers, Breast Density And Risk Reduction Perspectives In BRCA Carriers
Brief Title: Deslorelin Combined With Low-Dose Add-Back Estradiol and Testosterone in Preventing Breast Cancer in Premenopausal Women Who Are at High Risk for This Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 02164; P30CA033572 (NIH); CHNMC-IRB-02164; CDR0000355156 (Registry Identifier: NCI PDQ); NCI-2011-00975 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: brca1 Mutation Carrier; brca2 Mutation Carrier; Breast Cancer
Keywords: breast cancer; BRCA1 mutation carrier; BRCA2 mutation carrier
MeSH Terms: conditions — Breast Neoplasms | interventions — Estradiol; deslorelin; Testosterone Propionate; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (planned risk reduction mastectomy) (Experimental): Patients receive deslorelin, estradiol, and testosterone intranasally QD for 6 months. Patients then undergo planned risk reduction mastectomy.
  Interventions: Biological: therapeutic estradiol; Drug: deslorelin; Drug: therapeutic testosterone; Procedure: therapeutic conventional surgery; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis
- Group 2 (continued survaillance) (Active Comparator): Patients receive deslorelin, estradiol, and testosterone intranasally QD for 10 months. Patients then undergo continued surveillance through 10 months.
  Interventions: Biological: therapeutic estradiol; Drug: deslorelin; Drug: therapeutic testosterone; Other: active surveillance; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: therapeutic estradiol — 0.35mg/100ul per day as a nasal spray
Drug: deslorelin — 1mg/100ul per day as a nasal spray
Drug: therapeutic testosterone — 0.275mg/100ul per day as a nasal spray
Procedure: therapeutic conventional surgery — Undergo risk reduction mastectomy
  Arms: Group 1 (planned risk reduction mastectomy)
Other: active surveillance — Undergo continued surveillance
  Arms: Group 2 (continued survaillance)
Procedure: quality-of-life assessment — Ancillary studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Deslorelin combined with low-dose add-back estradiol and testosterone (given to replace hormones suppressed by deslorelin) may be effective in preventing breast cancer in at-risk women.

PURPOSE: This phase II trial is studying how well giving deslorelin together with estradiol and testosterone works in preventing breast cancer in premenopausal women who are at high risk for this disease.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Assess the effects on the breast of treatment with the gonadotropin-releasing hormone agonist (GnRHA)-based regimen in breast cancer (BRCA) gene mutation carriers, including correlation of changes in mammographic and magnetic resonance imaging (MRI) densities with tissue morphometrics and biomarkers.

II. Evaluate perspectives about risk reduction options and impact on quality-of-life (QOL) measures of participation in the chemopreventive protocol and in risk reduction surgery.

OUTLINE:

GROUP 1: Patients receive deslorelin, estradiol, and testosterone intranasally once daily (QD) for 6 months. Patients then undergo planned risk reduction mastectomy.

GROUP 2: Patients receive deslorelin, estradiol, and testosterone intranasally QD for 10 months. Patients then undergo continued surveillance through 10 months.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must generally be in good health with lab values and physical examination within normal limits
* Known high risk of breast cancer due to BRCA mutation or empiric risk > 30% lifetime by the Claus model
* No evidence or history of pervious cancer, except non-melanoma skin cancer
* Premenopausal women planning risk reduction mastectomy in 6 months or more (Group 1) or continued surveillance (Group 2)
* Prior tubal ligation or willing to use a non-hormonal barrier method of contraception
* Signed the Informed Consent Form document for this study in accordance with all Federal, State and Institutional regulations
* Must be current non-smoker

Exclusion Criteria:

* GnRHA treatment within 12 months of study entry
* Nasal polyposis, atrophic rhinitis, severe allergic or vasomotor rhinitis, or sinusitis requiring current treatment or treatment for more than 3 months in the previous year
* Concurrent medications including: corticosteroids (prednisone, prednisolone, cortisone acetate, Decadron, Deltasone, hydrocortisone, Hydrocortone, Medrol), estrogens, progestins or androgens, including oral, implanted, or injected contraceptive; (At least 6 months must have elapsed since the last use of an implanted or injected contraceptive such as Norplant)
* Pregnant or breast-feeding or have been so in the last six months
* Immeasurable breast density on mammogram

Ages: 21 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2004-03-11 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Treatment effects and correlation of changes in morphometrics and biomarkers as assessed by mammogram and magnetic resonance image (MRI) densities on days 1 and 300 | Day 300
Perspectives about risk reduction options and their impact on quality of life (QOL) as assessed by Medical Outcomes 36-item short-form version, Health Perceptions scale, and Body Image scale on days 1, 169, and 300, and then every 6 months for 2 years | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weitzel, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States